CLINICAL TRIAL: NCT02168582
Title: Improvement After Physiotherapy for Low Back Pain: The Good Responders. An Observational Study in Primary Care
Brief Title: Improvement After Physiotherapy for Low Back Pain: The Good Responders
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Trondheim Kommune (Other)
Responsible Party: Sponsor
Other Study IDs: LBP2014
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain
Keywords: Physical Therapy Modalities; Prognosis; Patient Selection
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities; Primary Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- low back pain
  Interventions: Behavioral: physiotherapy as usual in primary care

INTERVENTIONS:
Behavioral: physiotherapy as usual in primary care

SUMMARY:
This is an observational study that aims to characterize individual response of patients getting physical therapy for chronic non-specific low back pain.

Participants will be classified based on a questionnaire and motor tests to investigate whether individual improvement after physical therapy may be predicted. These observations may help to decide which should be the preferred treatment offered.

ELIGIBILITY:
Inclusion Criteria:

* low back pain
* receiving primary care physiotherapy

Exclusion Criteria:

-

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons seeking primary care physiotherapy because of low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
patient-reported disability | 1 year
  questionnaire (Oswestry Disability Index)

SECONDARY OUTCOMES:
self-efficacy | 1 year
  questionnaire and interview
global perceived effect | 1 year
  questionnaire
quality of life | 1 year
  questionnaire (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, prof md, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Public Health and General Practice, Trondheim, Norway